CLINICAL TRIAL: NCT06193278
Title: Personalized Neuromodulation Treatment for Parkinson's Syndrome
Brief Title: Individual Neuromodulation for PDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDS
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-08

CONDITIONS: Neuromodulation; Parkinsonian Syndromes; Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Parkinsonian Disorders | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- muti-site stimulation group1 (Active Comparator): The intervention period: 2 weeks muti-site: individual target (iTBS OR cTBS) / M1 (iTBS)
  Interventions: Device: Neuromodulation
- single-site stimulation group2 (Active Comparator): The intervention period: 2 weeks muti-site: individual target (sham) / M1 (iTBS)
  Interventions: Device: Neuromodulation
- sham stimulation group3 (Sham Comparator): The intervention period: 2 weeks muti-site: individual target (sham) / M1 (sham)
  Interventions: Device: Neuromodulation

INTERVENTIONS:
Device: Neuromodulation — Noninvasive brain stimulation (NIBS) includes a variety of noninvasive neuromodulation techniques such as transcranial magnetic stimulation (TMS), transcranial direct current stimulation (TDCS), and so on. Theta burst stimulation(TBS) is a new form of excitatory or inhibitory rTMS treatment that is less time-consuming and more effective than traditional rTMS in a single treatment session.

SUMMARY:
Parkinsonian Syndromes (PDS) with predominant motor dysfunction include progressive supranuclear palsy (PSP), multiple system atrophy (MSA) and corticobasal degeneration (CBD). Current treatment options for PDS are extremely limited due to the less understanding of disease pathophysiology and lack of therapeutic targets. Combining the results of previous studies and our group's previous research, sixty qualified PDS patients would be enrolled to conduct a prospective single-center randomized sham controlled clinical trial to verify the new therapeutic options that can improve symptoms and effectively slow the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with the MDS revised clinical diagnostic criteria for Parkinsonian syndrome (2015 edition)
* aged >40 years and <80 years, regardless of gender.
* Patients were relatively stable during the study period and remained stable on medication
* Good compliance, written informed consent, and consent for NIBS long-term intervention treatment

Exclusion Criteria:

* Patients with severe neuropsychiatric disorders or a previous history of severe neurologic conditions (e.g., epilepsy, cerebrovascular accident, etc.) or traumatic brain injury or brain surgery
* inability to complete the questionnaire independently
* Previous treatment with DBS or SCS; TMS or tDCS within 6 months
* Severe physical illness and any physical condition that can precipitate epilepsy or intracranial hypertension, including cardiovascular and respiratory diseases
* Installation of intracranial stents, pacemakers, coronary stents, cochlear implants, and other human implantable materials
* is currently taking other investigational drugs or is participating in other clinical trials
* Any other condition that the investigator believes makes him or her unsuitable for participation in this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Group differences of part 3 of Unified Parkinson Disease Rating Scale (UPDRS) changes | 6 weeks
  Compare the changes in UPDRS scores from baseline to post- treatment in the three intervention groups (UPDRS part3: range 0~72, higher score is related to a worse outcome).

SECONDARY OUTCOMES:
Group differences of Progressive Supranuclear Palsy Rating Scale (PSPRS) | 6 weeks
  Compare the changes in PSPRS scores from baseline to post- treatment in the three intervention groups (psp patients specific).
Group differences of Unified Multiple System Atrophy Rating Scale (UMSARS) | 6 weeks
  Compare the changes in UMSARS scores from baseline to post- treatment in the three intervention groups (MSA patients specific).
Group differences of Cortical Basal ganglia Functional Scale (CBFS) | 6 weeks
  Compare the changes in CBFS scores from baseline to post- treatment in the three intervention groups (cbd patients specific).
Group differences of Berg Balance Scale (BBS) changes | 6 weeks
  Compare the changes in BBS scores from baseline to post-treatment in the three intervention groups (BBS: range 0~56, higher score is related to a better outcome).
Group differences of Hamilton depression scale-17 (HAMD-17) changes | 6 weeks
  Compare the changes in HAMD-17 scores from baseline to post-treatment in the three intervention groups (HAMD-17: range 0~38, higher score is related to a worse outcome).
Group differences of Hamilton Anxiety Scale (HAMA) changes | 6 weeks
  Compare the changes in HAMA scores from baseline to post-treatment in the three intervention groups (HAMA: range 0~64, higher score is related to a worse outcome).
Group differences of Mini-mental State Examination (MMSE) changes | 6 weeks
  Compare the changes in MMSE scores from baseline to post-treatment in the three intervention groups (MMSE: range 0~30, higher score is related to a better outcome).
Group differences of Montreal Cognitive Assessment (MoCA) changes | 6 weeks
  Compare the changes in MoCA scores from baseline to post-treatment in the three intervention groups (MoCA: range 0~30, higher score is related to a better outcome).
Group differences of 39-item Parkinson's Disease Questionnaire (PDQ-39) changes | 6 weeks
  Compare the changes in PDQ-39 scores from baseline to post-treatment in the three intervention groups (PDQ-39: range 0~156, higher score is related to a worse outcome).
Group differences of Wexner scores changes | 6 weeks
  Compare the changes in Wexner scores from baseline to post-treatment in the three intervention groups (Wexner: range 0~30, higher score is related to a worse outcome).
Group differences of Standardized Swallowing Assessment (SSA) changes | 6 weeks
  Compare the changes in SSA from baseline to post-treatment in the three intervention groups
Group differences of adverse event | 6 weeks
  Compare the changes in adverse event in the three intervention groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology and Institute of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No